CLINICAL TRIAL: NCT00252538
Title: Genetic and Biochemical Markers of Interferon-Induced Depression.
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: MHBA-020-04F
Record Dates: First submitted 2005-11-09; First posted 2005-11-11 (Estimated); Results first posted 2014-12-11 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Depression
Keywords: Cortisol; Depression; Hepatitis C; Interferon; Polymorphism; Serotonin; Tryptophan
MeSH Terms: conditions — Depression; Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples are being collected to determine the variability in the development of depressive symptoms induced by interferon. Thus, we plan to measure specific genetic polymorphisms [i.e., in the serotonin (5-HT) transporter gene-linked polymorphic region (5-HTTLPR), in the promoter of the 5-HT1A receptor subtype, and an intronic tryptophan hydroxylase polymorphism]. Tryptophan, 5-HT, and cortisol blood levels will also be measured.

GROUPS / COHORTS (1):
- Group 1: Research participants are: 1) male or female, 2) age 18 or older, 3) chronically infected with the hepatitis C virus, 4) candidates for interferon therapy, 4) not on antidepressant treatment , and 5) not currently abusing any substances such as alcohol or intravenous drugs, or having abused in the past 6 months

SUMMARY:
The purpose of this study is to identify predictors and associated biochemical markers of interferon-induced depression. It is hypothesized that genetic variation in genes related to the serotonergic system may predict vulnerability to interferon-induced depression.

DETAILED DESCRIPTION:
1. Objective of project: Interferon-a (IFN)-induced depression is a common complication of its use in treating patients for hepatitis C (HCV), with reports of up to 44% of patients experiencing these depressive side effects. The central hypothesis of the proposed research is that polymorphisms in specific serotonergic genes are associated with a propensity to develop IFN-induced depression. Further, IFN-induced decreases in tryptophan and serotonin levels are putatively related to the emergence of depressive symptoms during IFN therapy. The objective of this proposal is to identify predictors of IFN-induced depression such that depressive side effects can be better managed and treated thus permitting patients to complete a full course of IFN therapy.
2. Research plan: We plan to test our hypothesis and accomplish the objectives of this application by pursuing the following two specific objectives:

   1. to evaluate the role of genetic loci that may contribute to the vulnerability to IFN using association analyses. Vulnerability is operationalized as the maximal Beck Depression Inventory-II (BDI-II) score, co-varying for pre-treatment BDI-II scores, and
   2. to identify the effects and time course of antiviral therapy on potential biomarkers of IFN-induced depression, including tryptophan, 5-HT, and cortisol levels. Changes in biochemical levels will be compared to depressive symptomology and genetic vulnerability.
3. Methodology: Patients will be asked to participate in a prospective study in which they will be monitored during the course of IFN therapy for symptoms of depression and for biochemical changes measured in their blood. 120 HCV patients initiating IFN therapy will be recruited (3/month for 40 months) from the Portland VA and the Long Beach VA Medical Centers. Following baseline assessments, subjects will be followed every 2 weeks for a period of 4 months. The development of major depression, depressive symptoms, and related IFN-induced side effects will be monitored using rating scales. For genetic and biochemical measures, blood samples will be collected prior to and during IFN therapy. Patients will be tested for certain genetic polymorphisms.

   Analyses. Using linear regression, genotype will be the independent variable, and co-varying for baseline BDI-II score, the maximal BDI-II score will be examined as a dependent variable. An ANOVA for repeated measures will be performed to determine the effects of IFN therapy on tryptophan, 5-HT, and cortisol levels. In addition, the relationship between interferon induced MDD and certain polymorphisms will be examined.
4. Findings, results or conclusions reached to date: In preliminary studies we found that 33% of HCV patients on IFN therapy developed major depressive disorder during the course of treatment. In addition, preliminary pilot results suggest that the 5-HT transporter polymorphism short allele and the "C" allele for the tryptophan hydroxylase polymorphism may increase vulnerability to IFN-induced depression.
5. Clinical relevance: There are currently no known, reliable predictors of IFN-induced depression. The chronic disease of HCV infection collectively affects approximately 4 million Americans and 200 million people worldwide. IFN is the only clinically approved medication whose long-term use can reduce the risk of a fatal outcome and even be curative in some individuals. However, side effects associated with IFN therapy represent a major obstacle to adequate treatment for patients with HCV, often resulting in the discontinuation IFN therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Serum positive for hepatitis C
2. Age 18 or older
3. Not pregnant and using adequate contraception
4. Hepatologist-determined patient is a candidate for interferon therapy
5. Written/signed informed consent specific for this protocol has been obtained prior to entry

Exclusion Criteria:

1. Diagnosis of active: depression, psychotic symptoms, or bipolar disorder (or history of bipolar disorder) during the previous 3 months
2. On antidepressant medications for any reason
3. Currently abusing any substances such as alcohol or intravenous drugs, or having abused in the past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 120 patients initiating interferon therapy will be recruited from the Portland, Minneapolis, and Long Beach VAMCs. The study is limited to only those participants who are currently mentally healthy at baseline and eligible to receive interferon therapy. Research participants are: 1) male or female, 2) age 18 or older, 3) chronically infected with the hepatitis C virus, 4) candidates for interferon therapy, 4) not on antidepressant treatment , and 5) not currently abusing any substances such as alcohol or intravenous drugs, or having abused in the past 6 months
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2006-04; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hauser, MD, Principal Investigator — VA Medical Center, Long Beach
Locations (3):
- United States (3):
  - VA Medical Center, Long Beach, Long Beach, California
  - VA Medical Center, Minneapolis, Minneapolis, Minnesota
  - VA Medical Center, Portland, Portland, Oregon

REFERENCES:
- [Result] Loftis JM, Patterson AL, Wilhelm CJ, McNett H, Morasco BJ, Huckans M, Morgan T, Saperstein S, Asghar A, Hauser P. Vulnerability to somatic symptoms of depression during interferon-alpha therapy for hepatitis C: a 16-week prospective study. J Psychosom Res. 2013 Jan;74(1):57-63. doi: 10.1016/j.jpsychores.2012.10.012. Epub 2012 Nov 21. PMID 23272989
- [Result] Lotrich FE, Loftis JM, Ferrell RE, Rabinovitz M, Hauser P. IL28B polymorphism is associated with both side effects and clearance of hepatitis C during interferon-alpha therapy. J Interferon Cytokine Res. 2011 Mar;31(3):331-6. doi: 10.1089/jir.2010.0074. Epub 2010 Dec 6. PMID 21133812
- See also: The Veterans Affairs National Hepatitis C Web site provides information about viral hepatitis for health care providers inside and outside the VA system, Veterans, and the General Public. — http://www.hepatitis.va.gov/
- See also: This is the Center for Disease Control's (CDC) website that provides information about Hepatitis C. — http://www.cdc.gov/ncidod/diseases/hepatitis/c/
- See also: The official website for the American Liver Foundation, which provides educational information and other resources for people with hepatitis C. — http://www.liverfoundation.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 133 participants from non- VA and VA sites were included for the genetic analysis. Patients from VA sites were recruited through/ referred by the local hepatology clinics. Recruitment occured from 4/6/2006 to 9/1/2009. A second manuscript included VA participants only.
Pre-assignment Details: Exclusion Criteria:
  1. Diagnosis of active: depression, psychotic symptoms, or bipolar disorder (or history of bipolar disorder) during the previous 3 months
  2. On antidepressant medications for any reason
  3. Currently abusing any substances such as alcohol or intravenous drugs, or having abused in the past 6 months.
Groups:
- Group 1 MDD; Group 2 Non MDD: Research participants are: 1) male or female, 2) age 18 or older, 3) chronically infected with the hepatitis C virus (HCV), 4) candidates for interferon therapy, 4) not on antidepressant treatment , and 5) not currently abusing any substances such as alcohol or intravenous drugs, or having abused in the past 6 months
  This is an observational study that segregates patients who have HCV and are started on interferon alpha treatment into 2 groups based on whether they develop major depressive disorder (MDD) while on interferon alpha therapy for HCV and then examines genes that may confer risk for MDD development. group 1 MDD and group 2 no MDD
Period: Overall Study
Arm/Group | Group 1 MDD | Group 2 Non MDD
Started | 19 | 114
Completed | 19 | 114
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Research participants are: 1) male or female, 2) age 18 or older, 3) chronically infected with the hepatitis C virus, 4) candidates for interferon therapy, 4) not on antidepressant treatment , and 5) not currently abusing any substances such as alcohol or intravenous drugs, or having abused in the past 6 months
  interferon-alpha: This is an observational study only. The patients are on interferon alpha therapy for HCV, but prescribing interferon is not a part of this research study protocol.
Arm/Group | Group 1
Number analyzed (Participants) | 133
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.1 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 100
Region of Enrollment [Number; unit: participants]
  United States | 133

OUTCOME MEASURES:

1. Primary Outcome: Phenotype and Genotype Based on Presence of Interferon Induced MDD.
Description: Structured psychiatric interviews and symptom rating scales for depression were used as primary outcome measures to determine the association between phenotype (interferon-induced depression) and genotype (genes that confer risk of interferon-induced depression). Genes of interest related to development of depression and antiviral treatment response that may confer risk for interferon induced depression were examined. this was a multi-site study and included participants from several hospital settings.
  Three polymorphisms of the interleukin (IL)-28b gene were examined - the c/c, c/t and t/t - and the relationship to MDD was examined. P-values above 0.05 are considered statistically insignificant in this study.
  In a subsequent analysis of only VA participants proinflammatory cytokines and serotonin levels were examined relative to symptoms of depression.
Time Frame: The proposed enrollment began after funding notification and enrollment will last for a period of 40 months and until end of study.
Population: This is an observational study that segregates patients with HCV and on interferon alpha treatment into 2 groups based on whether they develop major depressive disorder (MDD) while on interferon alpha therapy for HCV and then examines genes that may confer risk for MDD development. group 1 MDD and group 2 no MDD. total sample from multiple sites.
Measure: Number; unit: participants
Groups:
- Group 1- MDD; Group 2- no MDD: Research participants are: 1) male or female, 2) age 18 or older, 3) chronically infected with the hepatitis C virus, 4) candidates for interferon therapy, 4) not on antidepressant treatment , and 5) not currently abusing any substances such as alcohol or intravenous drugs, or having abused in the past 6 months
  This is an observational study that segregates patients who have HCV and are started on interferon alpha treatment into 2 groups based on whether they develop major depressive disorder (MDD) while on interferon alpha therapy for HCV and then examines genes that may confer risk for MDD development. group 1 MDD and group 2 no MDD
Arm/Group | Group 1- MDD | Group 2- no MDD
Number analyzed (Participants) | 19 | 114
participants | 19 | 114
Statistical Analysis 1: Comparison: Group 1- MDD vs Group 2- no MDD; All statistics employed Statistical Package for Social Science (SPSS) 17.0. Analysis of variances were used to compare viral responses in genotypes of interest, employing Scheffe's post-hoc analyses. Repeated-measure mixed-effect analyses were used to compare changes in subjective symptoms over time, including age, gender, and self identified race as covariates. Kaplan-Meier survival analyses examining time until MDD development were compared using theMantel-Cox log rank test; Test type: Superiority or Other; p > 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: 4/6/2006 - 9/1/2009 ( 3 years and 5 months)
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 1/133
Other Adverse Events (participants affected / at risk) | 0/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=133)
Elevation of Alpha Fetoprotein (Gastrointestinal disorders) | 1 (1) — Subject stopped Peginterferon and Ribavirin treatment. Patient was a non-responder to the treatment and also had an elevation of Alpha fetoprotein. A liver mass was detected in CT scan.

LIMITATIONS AND CAVEATS:
Limitations include that there are numerous polymorphism in various genes that may influence certain symptoms of depression. The risk for side effects during interferon-alpha treatment likely influenced by many genetic polymorphisms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes